CLINICAL TRIAL: NCT03580824
Title: A Phase 1b, Open-label, Age De-escalation, Dose-escalation Study to Evaluate the Safety and Immunogenicity of Different Doses of a Candidate Malaria Vaccine; Adjuvanted R21(R21/MM) in Adults, Young Children and Infants in Kilifi, Kenya
Brief Title: A Study to Determine if a New Malaria Vaccine is Safe and Induces Immunity Among Kenyan Adults, Young Children and Infants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Kenya Medical Research Institute (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VAC073
Record Dates: First submitted 2018-06-11; First posted 2018-07-09 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2022-08

CONDITIONS: Malaria,Falciparum
MeSH Terms: conditions — Malaria, Falciparum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Group 1 adults (n=20) will be administered 10mcg R21/50mcg Matrix-M vaccine through intramuscular route (into the non-dominant arm). A booster dose will be administered at 9-25 months post 3rd dose.
  Interventions: Biological: R21 in Matrix- M adjuvant vaccine
- Group 2 (Experimental): Group 2A children 1-5 years (n=3) will be receiving 5mcg R21/25mcg Matrix-M vaccine through intramuscular route (into the left deltoid).
  Group 2B children 1-5 years (n=17) will be receiving 10mcg R21/50mcg Matrix-M vaccine through intramuscular route (into the left deltoid). A booster dose will be administered at 9-25 months post 3rd dose.
  Interventions: Biological: R21 in Matrix- M adjuvant vaccine
- Group 3 (Experimental): Group 3A infants 5-<12 months (n=3) will be receiving 5mcg R21/25mcg Matrix-M vaccine through intramuscular route (into the left deltoid).
  Group 3B infants 5-<12 months (n=3) will be receiving 10mcg R21/50mcg Matrix-M vaccine through intramuscular route (into the left deltoid).
  Group 3C infants 5-<12 months (n=15) will be receiving 5mcg R21/25mcg Matrix-M vaccine through intramuscular route (into the left deltoid).
  Group 3D infants 5-<12 months (n=15) will be receiving 10mcg R21/50mcg Matrix-M vaccine through intramuscular route (into the left deltoid).
  Group 3E infants 5-<12 months (n=15) will be receiving 5mcg R21/50mcg Matrix-M vaccine through intramuscular route (into the left deltoid).
  A booster dose will be administered at 9-25 months post 3rd dose.
  Interventions: Biological: R21 in Matrix- M adjuvant vaccine

INTERVENTIONS:
Biological: R21 in Matrix- M adjuvant vaccine — R21: Protein particle malaria vaccine candidate in Matrix-M: Saponin based vaccine adjuvant.

SUMMARY:
This is a clinical trial to evaluate the safety and immunogenicity of R21/MM in healthy Kenyan participants from the different age groups.Participants will receive 3 vaccinations 4 weeks apart.

DETAILED DESCRIPTION:
The study includes three age groups:

Group 1: healthy adults (18-45 years) Group 2: young children (aged 1-5 years) Group 3: infants (aged 5- <12 months of age) Each group will receive 3 vaccine doses which will be 4-weeks apart. A booster dose will be administered at 9-25 months post 3rd dose.

The trial is funded by The European & Developing Countries Clinical Trials Partnership (EDCTP), European Union, ref: RIA2016V-1649 MMVC

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 45 years (Group 1), Healthy child aged 1-5 years (Group 2), healthy infant aged 5- <12 months (Group 3)
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Non-pregnant, non-lactating adult female or adult male
* Agreement to refrain from blood donation during the study
* Use of effective method of contraception for duration of study for female participants.

For female participants, we will ask them to attend with their family planning records for verification. Effective contraception is defined as a contraceptive method with failure rate of less than 1% per year when used consistently and correctly, in accordance with the product label. Examples of these include: combined oral contraceptives; injectable progestogen; implants of etenogestrel or levonorgestrel; intrauterine device or intrauterine system; male partner sterilisation at least 6 months prior to the female subject's entry into the study, and the relationship is monogamous; male condom combined with a vaginal spermicide (foam, gel, film, cream or suppository); and male condom combined with a female diaphragm, either with or without a vaginal spermicide (foam, gel, film, cream, or suppository)

* Adults with a Body Mass Index (BMI) 18 to 30 Kg/m2; or young children and infants with Z-score of weight-for-age within ±2SD
* Provide written informed consent
* Plan to remain resident in the study area for 2 years following last dose of vaccination

Exclusion Criteria:

* Clinically significant congenital abnormalities as judged by the study clinician.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (inhaled and topical steroids are allowed).
* Sickle cell trait or disease or G6PD deficiency.
* Any history of anaphylaxis in relation to vaccination.
* Clinically significant laboratory abnormality as judged by the study clinician.
* Blood transfusion within one month of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
* Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period.
* Seropositive for hepatitis B surface antigen (HBsAg) or hepatitis C (HCV IgG).
* Any significant disease, disorder or situation which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Ages: 5 Months to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 91 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of R21 with adjuvant Matrix-M in healthy adults then children and finally infants. | up to 2 years following vaccination
  Solicited and unsolicited adverse event data will be collected at each clinic visit from diary cards, clinical review, clinical examination (including observations) and laboratory results. This AE data will be tabulated and frequency, duration and severity of AEs compared between groups.
  The following parameters will be assessed for all study groups:
  * Occurrence of solicited local reactogenicity signs and symptoms for 7 days following the vaccination
  * Occurrence of solicited systemic reactogenicity signs and symptoms for 7 days following the vaccination
  * Occurrence of unsolicited adverse events for 28 days following the vaccination
  * Change from baseline for safety laboratory measures
  * Occurrence of serious adverse events during the whole study duration

SECONDARY OUTCOMES:
To assess the cellular and humoral immunogenicity of R21 in humans with adjuvant Matrix- M in healthy adults, children and infants. | up to 2 years following vaccination
  Comparison of immunogenicity (antibody responses) of the R21-Matrix-M1 - adjuvanted vaccination doses and the longevity of responses.
  * ELISA to quantify antibodies to the vaccine components CS, NANP and HBsAb.
  * Flow cytometry assays with intracellular cytokine staining to enumerate and functionally characterise immune cell populations such as effector and memory T cells (e.g. CD4+ and CD8+), T follicular helper cells, regulatory T cells, B cells, plasma cells and dendritic cells
  * ELISPOT for enumeration of antibody-secreting cells (e.g. B and plasma cells)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hill, Principal Investigator — University of Oxford
Locations (1):
- KEMRI/Wellcome Trust Programme, Centre for Geographic Medicine Research - Coast, Kilifi, Kenya

REFERENCES:
- [Derived] Mukhopadhyay ES, Bellamy DG, Tinto H, Hamaluba M, Truby A, Salman AM, Hill AVS. Naturally acquired immune responses to alpha-gal in malaria endemic settings and pre-clinical efficacy testing with R21/MM. Vaccine. 2025 Dec 5;68:127897. doi: 10.1016/j.vaccine.2025.127897. Epub 2025 Nov 1. PMID 41176969
- [Derived] Sang S, Datoo MS, Otieno E, Muiruri C, Bellamy D, Gathuri E, Ngoto O, Musembi J, Provstgaard-Morys S, Stockdale L, Aboagye J, Woods D, Lawrie A, Roberts R, Keter K, Kimani D, Ndungu F, Kapulu M, Njau I, Orindi B, Ewer KJ, Hill AVS, Bejon P, Hamaluba M. Safety and immunogenicity of varied doses of R21/Matrix-M vaccine at three years follow-up: A phase 1b age de-escalation, dose-escalation trial in adults, children, and infants in Kilifi-Kenya. Wellcome Open Res. 2023 Oct 12;8:450. doi: 10.12688/wellcomeopenres.19795.1. eCollection 2023. PMID 38813551